CLINICAL TRIAL: NCT00660504
Title: Randomized, Open-label, phase3 Trial Comparing Amrubicin Combined With Cisplatin Versus Etoposide-Cisplatin as First-line Treatment in Patients With Extensive Disease SCLC
Brief Title: Phase3 Study of Amrubicin With Cisplatin Versus Etoposide-cisplatin for Extensive Disease Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0750018; D0750018
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Lung Cancer
Keywords: Extensive Disease-Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Amrubicin Hydrochloride-Cisplatin combined chemotherapy
  Interventions: Drug: Amrubicin Hydrochloride
- 2 (Active Comparator): Etoposide-Cisplatin combined chemotherapy
  Interventions: Drug: Etoposide-Cisplatin combined chemotherapy

INTERVENTIONS:
Drug: Amrubicin Hydrochloride — Amrubicin Hydrochloride combined with cisplatin
  Arms: 1
Drug: Etoposide-Cisplatin combined chemotherapy — combined chemotherapy
  Arms: 2

SUMMARY:
This study drug(Amrubicin)is believed to work by stopping the tumor cell in your body from growing. The purpose of this study is to evaluate the efficacy and safety of amrubicin with cisplatin compared to etoposide-cisplatin in the first-line treatment in extensive disease small cell lung cancer The subject, who is randomized to AP group may be involved into a pharmacokinetic study of amrubicin and the metabolites: amrubicinol voluntarily.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically proven small cell lung cancer
* Extensive disease
* No prior chemotherapy regimen
* Age 18 years or older
* ECOG performance status of 0-1

Exclusion Criteria:

* Brain metastasis requiring treatment
* Treatment (Surgical or radiotherapy)of primary tumor
* Interstitial pneumonia or pulmonary fibrosis
* Abnormal cardiac function or myocardial infraction within 6 months before study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-04; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Sun, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (15):
- China (15):
  - Fuzhou, Fujian
  - Lanzhou, Gansu
  - Guangzhou, Guangdong
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Nanchang, Jiangxi
  - Changchun, Jilin
  - Dalian/Shenyang, Liaoning
  - Shenyang, Liaoning
  - Xian, Shanxi
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai
  - Tianjin

REFERENCES:
- [Derived] Sun Y, Cheng Y, Hao X, Wang J, Hu C, Han B, Liu X, Zhang L, Wan H, Xia Z, Liu Y, Li W, Hou M, Zhang H, Xiu Q, Zhu Y, Feng J, Qin S, Luo X. Randomized phase III trial of amrubicin/cisplatin versus etoposide/cisplatin as first-line treatment for extensive small-cell lung cancer. BMC Cancer. 2016 Apr 9;16:265. doi: 10.1186/s12885-016-2301-6. PMID 27061082

RESULTS

PARTICIPANT FLOW:
Groups:
- Amrubicin Combined With Cisplatin Group: Amrubicin Hydrochloride-Cisplatin combined chemotherapy
  Amrubicin Hydrochloride : Amrubicin Hydrochloride combined with cisplatin
- Etoposide Combined With Cisplatin Group: Etoposide-Cisplatin combined chemotherapy
  Etoposide-Cisplatin combined chemotherapy : combined chemotherapy
Period: Overall Study
Arm/Group | Amrubicin Combined With Cisplatin Group | Etoposide Combined With Cisplatin Group
Started | 149 | 151
Completed | 149 | 150
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amrubicin, Anticancer, Injection | Etoposide, Anticancer, Injection | Total
Number analyzed (Participants) | 149 | 150 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (10.03) | 57.45 (9.78) | 56.78 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 114 | 113 | 227
Region of Enrollment [Number; unit: participants]
  China | 149 | 150 | 299

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: 1.5 years after last subject enrolled
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Amrubicin Combined With Cisplatin Group | Etoposide Combined With Cisplatin Group
Number analyzed (Participants) | 149 | 150
month | 11.79 [11.01 to 12.62] | 10.28 [9.23 to 11.96]

2. Other Pre Specified Outcome: Overall Survival at 6 and 12 Months
Time Frame: 6 and 12 months.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Amrubicin Combined With Cisplatin Group | Etoposide Combined With Cisplatin Group
Number analyzed (Participants) | 149 | 150
percentage of patients
  6-month | 89.26 [83.07 to 93.28] | 86.00 [79.34 to 90.64]
  12-month | 48.59 [40.31 to 56.36] | 41.93 [33.97 to 49.68]

3. Secondary Outcome: Progression-Free Survival
Time Frame: 1.5 years after last subject enrolled
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Amrubicin Combined With Cisplatin Group | Etoposide Combined With Cisplatin Group
Number analyzed (Participants) | 149 | 150
month | 6.83 [6.11 to 7.39] | 5.72 [5.06 to 6.93]

4. Secondary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: participants were followed for the duration of the study, an average of 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Amrubicin Combined With Cisplatin Group | Etoposide Combined With Cisplatin Group
Number analyzed (Participants) | 149 | 150
percentage of participants | 69.80 | 57.33

ADVERSE EVENTS:
Arm/Group | Amrubicin, Anticancer, Injection | Etoposide, Anticancer, Injection
Serious Adverse Events (participants affected / at risk) | 21/149 | 8/150
Other Adverse Events (participants affected / at risk) | 149/149 | 148/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amrubicin, Anticancer, Injection (N=149) | Etoposide, Anticancer, Injection (N=150)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia syndrome (Blood and lymphatic system disorders) | 3 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 5 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmias (Cardiac disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 | 0
fever (Infections and infestations) | 2 | 0
Chronic cholecystitis (Vascular disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Lower hemoglobin (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 7 | 0
Platelet count decreased (Investigations) | 3 | 1
White blood cell count decreased (Investigations) | 6 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2
Dyskinesia (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Acute renal failure (Renal and urinary disorders) | 1 | 0
Mental disorders (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amrubicin, Anticancer, Injection (N=149) | Etoposide, Anticancer, Injection (N=150)
Nausea (Gastrointestinal disorders) | 72 | 70
vomit (Gastrointestinal disorders) | 63 | 63
Decreased appetite (Gastrointestinal disorders) | 60 | 50
Constipation (Gastrointestinal disorders) | 32 | 25
Alopecia (General disorders) | 31 | 20
fever (Infections and infestations) | 28 | 12
Fatigue (General disorders) | 27 | 11
Diarrhea (Gastrointestinal disorders) | 25 | 13
Gastrointestinal Disorders (Gastrointestinal disorders) | 22 | 26
Neutrophil count decreased (Blood and lymphatic system disorders) | 99 | 85
White blood cell count decreased (Blood and lymphatic system disorders) | 97 | 85
Platelet count decreased (Blood and lymphatic system disorders) | 54 | 40
Lower hemoglobin (Blood and lymphatic system disorders) | 49 | 50
Anemia (Blood and lymphatic system disorders) | 48 | 48
Bone marrow failure (Blood and lymphatic system disorders) | 46 | 46
Decreased red blood cell count (Blood and lymphatic system disorders) | 14 | 15
Mouth ulcers (Gastrointestinal disorders) | 9 | 6
Abnormal liver function (Hepatobiliary disorders) | 8 | 5
Lymphocyte count decreased (Investigations) | 13 | 5
Reduced red blood cell count (Investigations) | 14 | 15
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 4
Hypochloraemia (Metabolism and nutrition disorders) | 9 | 2
Hypokalemia (Metabolism and nutrition disorders) | 13 | 6
Hyponatremia (Metabolism and nutrition disorders) | 12 | 5
Dizziness (Nervous system disorders) | 10 | 6
Headache (Nervous system disorders) | 9 | 1
Insomnia (Psychiatric disorders) | 11 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Hiccup (Respiratory, thoracic and mediastinal disorders) | 8 | 10
alanine aminotransferase increased (General disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days